CLINICAL TRIAL: NCT07126158
Title: Phase II Study of Stereotactic Body Radiotherapy Plus FAK and RAF/MEK Inhibition in Advanced Pancreatic Adenocarcinoma
Brief Title: Stereotactic Body Radiotherapy Plus FAK and RAF/MEK Inhibition in Advanced Pancreatic Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Verastem, Inc. (Industry); The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-x348
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Adenocarcinoma; Cancer of the Pancreas; Pancreas Cancer; Pancreatic Cancer
Keywords: Pancreas cancer; SBRT; FAK; MEK
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery; defactinib

STUDY DESIGN:
Intervention Model Description: Patients will be randomized on a 5:1 basis to the Experimental Arm or the Control arm. The first 6 patients randomized and treated on the Experimental Arm will be considered the safety lead-in. Following completion of the safety lead-in, additional patients will be accrued in order to reach a total of 30 patients on the Experimental arm (inclusive of the safety lead-in cohort) and 6 on the Control arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental Arm: SBRT + Defactinib + Avutometinib (Experimental): Participants will receive approximately 12 months of treatment on study with 5 fractions of adaptive SBRT with 12 cycles of oral defactinib + avutometinib beginning on Day 2 of radiation. Cycles are 28 days in length. Defactinib is dosed twice a day and avutometinib is dosed twice a week (e.g. Monday and Thursday, Tuesday and Friday, etc.) on a 3 weeks on, 1 week off schedule. The first 6 participants will be enrolled in the Safety Lead-In cohort to monitor for dose-limiting toxicities. Patients who are candidates for surgical resection will undergo standard of care surgery at 2 weeks post-end of SBRT (+/- 1 weeks) or 12 weeks post-end of SBRT (+/- 1 week). These patients will discontinue defactinib and avutometinib the day prior to the operation and will resume taking it 4 to 6 weeks after surgery for the remainder of the 12 cycles. Patients who are not candidates for surgical resection will continue to receive defactinib plus avutometinib uninterrupted.
  Interventions: Radiation: Stereotactic body radiotherapy; Drug: Defactinib; Drug: Avutometinib
- Control Arm: SBRT (Active Comparator): Participants will receive 5 fractions of adaptive SBRT.
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — MRIdian and Ethos (adaptive radiation platforms)
  Other Names: SBRT
Drug: Defactinib — Taken with 30 minutes of a meal
  Arms: Experimental Arm: SBRT + Defactinib + Avutometinib
Drug: Avutometinib — Can be taken without regard to food.
  Arms: Experimental Arm: SBRT + Defactinib + Avutometinib

SUMMARY:
Advanced pancreatic cancer patients receiving treatment of adaptive stereotactic body radiotherapy (SBRT) with concurrent and adjuvant defactinib plus avutometinib will have increased progression-free survival (PFS) compared to historical PFS rates for patients receiving adaptive SBRT alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced pancreatic adenocarcinoma that is considered borderline resectable or locally advanced per institutional standardized criteria of unresectability or medical inoperability (NCCN guidelines 2.2021 PANC-C 1 of 2).
* Patients with locoregional adenopathy are eligible as long as all suspicious lymph nodes are deemed to be adjacent to the primary tumor as per radiation oncologist assessment.
* Patients must have received at least 2 months of systemic chemotherapy for this disease without progression of local or systemic disease. Newly diagnosed patients may be screened for enrollment in this study and can be enrolled once they have completed 2 months of systemic chemotherapy (and still meet all eligibility criteria) prior to the start of study treatment.
* At least 18 years of age.
* ECOG performance status ≤ 1.
* Life expectancy > 3 months
* Adequate bone marrow and organ function within 21 days of C1D1 as defined below:

  * Absolute neutrophil count ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN; no prior history of Gilbert's syndrome
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN or ≤ 5.0 x IULN if due to liver involvement by tumor
  * Creatinine clearance ≤ 1.5 x IULN or glomerular filtration rate of ≥ 60 mL/min
  * INR ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of anticoagulants
  * aPTT ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of anticoagulants
  * Albumin ≥ 2.5 mg/dL
  * Creatine phosphokinase (CPK) ≤ 2.5 x IULN
* Adequate cardiac function with left ventricular ejection fraction ≥ 55% by echocardiography (ECHO) or multiple-gated acquisition (MUGA) scan.
* Corrected QT interval (QTc) < 480 ms (as calculated by the Fridericia correction formula).
* The effects of defactinib and avutometinib on the developing human fetus are unknown. For this reason and because radiation therapy is known to be teratogenic, women of childbearing potential and men must agree to use highly effective contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study and up to 30 days after completion of treatment, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and 90 days after completion of the study
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease.
* Clinically evident ascites or pleural effusion that requires therapeutic paracentesis or thoracentesis.
* Prior treatment with a drug of the FAK inhibitor or RAF/MEK inhibitor class, or with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte associated antigen 4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Prior anti-human antibody response (AHA or ADA).
* Currently receiving any other investigational agents or has received any other investigational agents within 4 weeks or 5 half-lives, whichever is shorter, of C1D1.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to defactinib, avutometinib, or other agents used in the study, or a history of hypersensitivity to any of the inactive ingredients (hydroxypropylmethylcellulose, mannitol, magnesium stearate) of the investigational product.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy not routinely associated with chemotherapeutic regimen.
* Requires continued use of warfarin for anticoagulation and cannot stop warfarin or be safely switched to another anticoagulant or direct oral anticoagulant.
* Has an active autoimmune disease requiring systemic treatment with use of disease modifying agents, corticosteroids, or immunosuppressive drugs within the past 2 years. Replacement therapy such as thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc. is not considered a form of systemic treatment.
* Received a live vaccine within 30 days prior to the first study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist) are live attenuated vaccines and are not allowed.
* Known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV RNA [qualitative] is detected).
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has a known history of active TB (bacillus tuberculosis).
* Major surgery within 28 days prior to the first study treatment.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.
* Known SARS-Cov2 infection ≤28 days prior to first dose of study therapy.
* Exposure to medications (with or without prescriptions), supplements, herbal remedies, or foods with potential for drug-drug interactions with avutometinib and/or defactinib within 5 half-lives (if half-life is known) or 14 days prior to C1D1. Specifically, this includes:

  * Strong CYP3A4 inhibitors or inducers
  * Strong CYP2C9 inhibitors or inducers
  * Strong P-glycoprotein (P-gp) inhibitors or inducers
  * Strong breast cancer resistance protein (BCRP) inhibitors or inducers.
* Subjects with the inability to swallow oral medications or impaired gastrointestinal absorption due to gastrectomy or active inflammatory bowel disease.
* Subjects with an active skin disorder that has required systemic therapy within the past year and may confound the interpretation of the safety findings from the study treatments, in the opinion of the investigator.
* History of medically significant rhabdomyolysis.
* Patients with concurrent ocular disorders:

  * Patients with history of glaucoma, history of retinal vein occlusion (RVO), predisposing factors for RVO, including uncontrolled hypertension, uncontrolled diabetes.
  * Patients with history of retinal pathology or evidence of visible retinal pathology that is considered a risk factor for RVO, intraocular pressure > 21 mm Hg as measured by tonometry, or other significant ocular pathology, such as anatomical abnormalities that increase the risk for RVO.
  * Patients with active or chronic, visually significant corneal disorders, other active ocular conditions requiring ongoing therapy or clinically significant corneal disease that prevents adequate monitoring of drug-induced keratopathy. Examples of visually significant corneal disorders include corneal degeneration, active or recurrent keratitis, and other forms of serious ocular surface inflammatory conditions. Visually significant corneal disorders do NOT include dry eyes, blepharitis, and uncomplicated corneal erosions.
* Concurrent congestive heart failure, prior history of class III/ IV cardiac disease (New York Heart Association [NYHA]), myocardial infarction within the last 6 months, unstable arrhythmias, unstable angina or severe obstructive pulmonary disease.
* Any other medical condition (eg, cardiac, gastrointestinal [eg, severe heartburn, gastric ulcer, etc], pulmonary, psychiatric, neurological, genetic, GI bleeding, substance abuse, alcoholism, etc) within 3 months prior to enrollment that, in the opinion of the Investigator, would place the patient at unacceptably high risk for toxicity.
* Active, uncontrolled infection (bacterial, viral, or fungal) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment. Subjects must be afebrile for > 48 hours off systemic therapy.
* Symptomatic brain metastases requiring steroids or other local interventions. Patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study entry, have discontinued corticosteroid treatment for these metastases for at least 2 weeks prior to first dose of study therapy, and are neurologically stable, with no evidence of interim progression. Patients with new asymptomatic CNS metastases detected during the screening period must receive radiation therapy and/or surgery for CNS metastases. Following treatment, these patients may then be eligible if all other criteria are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) - Experimental Arm Only | Through completion of follow-up (up to 2 years)

SECONDARY OUTCOMES:
Number of patients with acute toxicity - Experimental Arm Only | From start of treatment through 90 days
  Graded by CTCAE v. 5.0
Number of patients with late toxicity - Experimental Arm Only | From day 91 through 2 years
  Graded by CTCAE v. 5.0
Local control - Experimental Arm Only | At 12 months
Distant metastasis progression-free survival (DM-PFS) - Experimental Arm Only | Through completion of follow-up (up to 2 years)
Objective response rate (ORR) - Experimental Arm Only | At 12 weeks post-adaptive SBRT (estimated to be 13 weeks)
Overall survival (OS) - Experimental Arm Only | Through completion of follow-up (up to 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Grierson, M., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu